CLINICAL TRIAL: NCT05799807
Title: Weight-bearing Diagnostics in Acute Lisfranc Injury: A Prospective Study Comparing Computed Tomography Versus Conventional Radiography
Brief Title: Weight-bearing Diagnostics in Acute Lisfranc Injury: CT vs X-ray
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Poulsen, Principal Investigator, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 110364
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Lisfranc Injury; Foot Sprain
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Acute Lisfranc injuries are investigated with weight-bearing diagnostics to determine the degree of TMT stability. Patients are examined using both CT and conventional radiography during full weight and non-weight-bearing sequences. 3 foot- and ankle surgeons will examine the scans independently, starting with the conventional radiographs. Distance between the medial cuneiform and second metatarsal bone (C1-M2) is measured. For the CT images, measuring method previously described by Y. Sripanich et al. (DOI: 10.1007/s00402-020-03477-5) will be used.
  CT findings will determine the treatment outcome. If the C1-M2 diastasis is >2mm, as opposed to the uninjured side, the injury will be determined unstable and surgical fixation will be recommended (Cohort 2). All other patients (≤ 2mm) are considered stable and treated conservatively (Cohort 1).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Conservative (Active Comparator): Negative weight-bearing CT (≤ 2mm between C1-M2, as opposed to the uninjured side) will be considered stable and treated conservatively with a prefabricated walker with weight-bearing as tolerated for six weeks. These patients will undergo bilateral radiographs after six weeks and combined CT and radiographs after twelve weeks to monitor the degree of stability
  Interventions: Procedure: Conservative treatment
- Cohort 2 - Surgical (Active Comparator): Positive weight-bearing CT (> 2mm between C1-M2, as opposed to the uninjured side) will be operated by minimally invasive stabilization (eg, isolated homerun screw)
  Interventions: Procedure: Minimally invasive stabilization

INTERVENTIONS:
Procedure: Conservative treatment — Patients with negativ weight-bearing CT will be treated conservative
  Arms: Cohort 1 - Conservative
Procedure: Minimally invasive stabilization — Patients with positive weight-bearing CT will be operated by minimally invasive stabilization (eg, isolated homerun screw)
  Arms: Cohort 2 - Surgical

SUMMARY:
A prospective, cohort study comparing weight-bearing computed tomography with weight-bearing radiography in patients with an acute Lisfranc injury.

DETAILED DESCRIPTION:
Injury to the tarsometatarsal (TMT) joint complex in the midfoot is referred to as a Lisfranc injury. The broad spectrum of these injuries includes simple sprains to severe fracture-dislocations. Variable clinical presentations and radiographic findings make Lisfranc injuries notoriously difficult to detect, especially in the case of subtle ligament injuries. Nowadays, up to 30% of unstable Lisfranc injuries are overlooked or misdiagnosed. This can potentially lead to severe sequelae such as post-traumatic osteoarthritis and foot deformities.

For obvious injuries involving diastasis, subluxation, or dislocation, the diagnosis is relatively easy to establish using any imaging modality. However, for subtle injuries without gross bone separation, a dynamic imaging modality facilitating weight-bearing are to be preferred. Many consider weight-bearing conventional radiography as the current gold standard in acute Lisfranc injury diagnostics. However, conventional radiography is a 2D technique that can neither display nor measure the true dimensions of a detailed 3D object, such as the tarsal bones in the foot. Computed tomography (CT) provides greater accuracy in visualizing bone microarchitecture. In combination with weight-bearing, it can be ideal for detecting minor fractures and occult instability caused by load/stress.

To this day, there are no prospective studies comparing weight-bearing CT and weight-bearing radiography for acute Lisfranc injuries. In the current study, participants will be assigned to non-operative or operative treatment based on Lisfranc joint stability evaluation by the initial weight-bearing CT.

ELIGIBILITY:
Inclusion Criteria:

* Acute trauma to the midfoot
* Intraarticular fracture and/or avulsion fracture in the TMT joint line (detected on a non-weight-bearing CT)
* Suspicion of a purely ligamentous Lisfranc injury (no radiological fractures but substantial clinical findings in the midfoot region, or evidence of ligamentous damage on a MRI)
* Consent-competent patient

Exclusion Criteria:

* Obvious acute unstable Lisfranc injuries (>2mm dislocation between the medial cuneiform and second metatarsal)
* Injury older than four weeks
* Other major foot/ankle/leg injuries
* Previous foot infection or foot pathology on the affected side
* Previous surgery to the TMT joints, and sequelae after a previous foot injury
* Open injury
* Bilateral injury
* Patients with co-morbidities such as neuropathy and peripheral vascular disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Manchester-Oxford Foot Questionnaire (MOxFQ) | 1 year
  Foot-Ankle specific PROM (0-100 with 0 representing the best possible outcome)

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Midfoot score | 1 year
  Foot-Ankle specific PROM (0-48 with 48 representing the best possible outcome)
Visual Analogue Scale (VAS) for pain | 1 year
  Scores pain at rest and on activity (0-10 with 0 representing no pain)
Short-Form (SF) 36 | 1 year
  Patient reported score measuring quality of life and health status (0-100 with 100 representing the best possible outcome)
Posttraumatic osteoarthritis | 1 year
  The presence of osteoarthritis of the tarsometatarsal joints using the Kellgren & Lawrence classification system
Incidence of complications | 1 year
  Yes/no for deep or superficial infection, nerve or tendon injury, deep venous thrombosis, hardware complaints and secondary surgery. Regards the patients that have undergone surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Poulsen, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No